CLINICAL TRIAL: NCT04849156
Title: Sperm Selection by Thermotaxis: a Novel Technique to Enhance Assisted Reproductive Technologies' Outcomes
Brief Title: Spermatozoa Morphology Selection by Thermotaxis
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidade de Lisboa (Network)
Responsible Party: Sponsor
Other Study IDs: 1902-LIS-028-SR
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Male Infertility
Keywords: Spermatozoa selection; Thermotaxis; Testicular and sperm biology
MeSH Terms: conditions — Infertility, Male; Taxis Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sperm samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sperm selection by thermotaxis — Selection of healthy sperm by thermotaxis procedure

SUMMARY:
This study aims to eventually assess the usefulness of thermotaxis for sperm selection in routine clinical practice.

DETAILED DESCRIPTION:
As the world's total fertility rate decline, every year more couples require assisted reproductive technologies (ART) in order to achieve their desire to become parents. However, these techniques are not guaranteed solutions and still many couples with unexplained infertility fail to conceive. One of the reasons might be the relative selection of spermatozoa for the following ART. To minimize a poor selection made by the operator and to standardize spermatozoa selection, we suggest a new method might be used in combination with the routine spermatozoa selection techniques.

Thermotaxis might be used in the ART setting as a tool to select the best spermatozoa as human spermatozoa after capacitation responds positively to a temperature gradient change. Moreover, this might be the possible navigation mechanism of spermatozoa in the female genital tract. We hypothesize that spermatozoa selected by thermotaxis behavior might increase the morphologically normal spermatozoa number in the cohort used during ART.

The aim of this study is to evaluate if thermotaxis is a good method for selecting morphologically normal sperm for ART.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 and <40 years old.
* Spermatozoa concentration >15 x 10⁶ /mL in all sperm analysis performed in the last 24 months.
* Spermatozoa mobility >32% in all sperm analysis performed in the last 24 months.
* Spermatozoa morphology >4% in all sperm analysis performed in the last 24 months.
* Signed and dated informed consent

Exclusion Criteria:

* Use of antibiotics, intravenous illicit drugs, chemotherapy or radiotherapy usage in the last 3 months.
* Active smoking (during the preceding 12 months).
* More than 3 days prior to the last ejaculation.

Ages: 18 Years to 39 Years | Sex: Male
Age Groups: Adult
Gender Based: Yes
Study Population: 10 male sperm donors.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Percentage of normal spermatozoa morphology | 11 months
  Analysis of sperm samples following thermotaxis (intervention) versus the controls (without thermotaxis).

CONTACTS AND LOCATIONS:
Overall Officials: Kadir Guleresi, Master, Principal Investigator — Instituto Valenciano de Infertilidade de Lisboa
Locations (1):
- Instituto Valenciano de Infertilidade de Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No